CLINICAL TRIAL: NCT01138020
Title: Cognitive Rehabilitation of Blast-induced Traumatic Brain Injury
Brief Title: Cognitive Rehabilitation of Blast Traumatic Brain Injury (TBI)
Acronym: CRbTBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6996-W
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury; Cognitive Symptoms
Keywords: Rehabilitation Outcome; Cognitive treatment; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurobehavioral Manifestations | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Cognitive intervention
  Interventions: Behavioral: Cognitive Intervention
- Arm 2 (Active Comparator): Educational intervention
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Cognitive Intervention — Cognitive rehabilitation treatment designed specifically to address the most common cognitive complaints in executive and memory function
  Arms: Arm 1
Behavioral: Educational intervention — Educational intervention is geared at personal management of TBI-related symptoms.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to investigate the efficacy of a structured rehabilitation program on cognitive function and quality of life in individuals with blast-induced traumatic brain injury (bTBI).

DETAILED DESCRIPTION:
The most common impairments following blast-induced traumatic brain injury (bTBI) are cognitive deficits in the domain of executive functioning, learning and memory, and functional and psychosocial disabilities that are closely related to these cognitive deficits. There are no treatment protocols available to address the multiple cognitive impairments in bTBI, but cognitive rehabilitation has proven efficacious in the treatment of non-blast TBI. The cognitive training modules the investigators plan to evaluate have improved organization and memory function in patients with non-blast TBI, but it is unknown whether their efficacy exceeds that of programs that focus only on education and support. This study is a between group comparison of a cognitive rehabilitation treatment designed specifically to address the most common cognitive complaints in executive and memory function, and an active control group receiving educational intervention geared at personal management of TBI-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) active-duty personnel or Veterans exposed to blast
* Meets criteria for mild TBI
* loss of consciousness (LOC) of 30 min or less
* Age: 21- 50

Exclusion Criteria:

* Evidence of penetrating head injury
* History of previous neurological diagnosis
* History of previous psychotic disorder prior to the blast exposure
* Hearing or vision impairment

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning | Ten weeks
  Scaled Score on the standardized neuropsychological testing

SECONDARY OUTCOMES:
Daily functioning | Ten weeks
  Total Score on the daily functioning measure

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Bogdanova, PhD PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No